CLINICAL TRIAL: NCT01914744
Title: Entecavir Versus Lamivudine for Preventing the Risk of Hepatitis B Virus Reactivation in Patients With Non-Hodgkin Lymphoma on CHOP/R-CHOP: a Randomized Phase II Study
Brief Title: Entecavir Versus Lamivudine for Preventing the Risk of Hepatitis B Reactivation in NHL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LMTG 13-03
Record Dates: First submitted 2013-03-02; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Non-Hodgkin Lymphoma; Hepatitis B Reactivation
Keywords: NHL; HBV; entecavir; lamivudine
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — entecavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- entecavir (Experimental): entecavir 0.5 mg/day PO
  Interventions: Drug: Entecavir; Drug: Lamivudine
- lamivudine (Active Comparator): lamivudine 100 mg/day PO
  Interventions: Drug: Entecavir; Drug: Lamivudine

INTERVENTIONS:
Drug: Entecavir — entecavir 0.5 mg/day PO
  Other Names: baraclude
Drug: Lamivudine — lamivudine 100 mg/day PO
  Other Names: epivir

SUMMARY:
The aim of this study is to prove the superiority of entecavir over lamivudine for preventing the risk of hepatitis B virus reactivation in patients with non-Hodgkin lymphoma on CHOP/R-CHOP.

DETAILED DESCRIPTION:
In china, previous studies showed patients with non-Hodgkin lymphoma (NHL) are likely to have hepatitis B virus (HBV) infection. The risk of HBV reactivation is high when patients were treated with CHOP, especially in combination with rituximab. The aim of this study is to compare entecavir with lamivudine, 2 commonly used anti-virus agents, for preventing the risk of HBV reactivation in patients with NHL on CHOP/R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated NHL suitable for CHOP/R-CHOP treatment
* Age range 18-80 years old
* HBsAg positive with high level of HBV DNA
* Eastern Cooperative Oncology Group performance status 0-2
* Life expectancy of more than 3 months
* Adequate organ function

Exclusion Criteria:

* Primary or secondary central nervous system involvement
* With hepatitis C virus infection
* Previous serious cardiac disease
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of HBV reactivation | 12 months
  Defined by increased level of HBV DNA

SECONDARY OUTCOMES:
Incidence rate of hepatitis and HBV reactivation-related hepatitis | 6 months
  Defined by increased level of alanine transaminase
Incidence rate and median time of treatment delay due to hepatitis | 6 months
  Measured by information of treatment delay
Incidence rate and median time of HBV DNA level normalization | 6 months
  Measured by information of HBV DNA level normalization

OTHER OUTCOMES:
Incidence of drug resistance of viral variants | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China